CLINICAL TRIAL: NCT07276126
Title: The Effect of the Cesarean ERAS Protocol on Mother-Infant and Father-Infant Bonding: a Multicenter, Randomized Controlled Clinical Trial.
Acronym: ERAS-CS-BOND-1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Responsible Party: Principal Investigator, Gökçenur Karakelleoğlu, Assisted Prof, Okan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-66291034-202.3.02-7579
Record Dates: First submitted 2025-11-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Bonding; ERAS; Cesarean Section; Maternal Care; Father - Child Relations; Mother-Infant Interaction
Keywords: eras; erac; cesarean; maternal bonding; paternal bonding

STUDY DESIGN:
Intervention Model Description: Arm 1: ERAS Protocol
  Arm 2: Standard Perioperative Care
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS Protocol (Active Comparator): Participants in this arm will receive the Enhanced Recovery After Cesarean (ERAS) protocol, which includes preoperative patient education and anxiety reduction, intraoperative multimodal analgesia, early oral intake, early mobilization, and early removal of Foley catheter. Skin-to-skin contact and early breastfeeding will be encouraged, and fathers will be actively involved in postpartum care. Outcomes include mother-infant and father-infant bonding, maternal postpartum depression, breastfeeding initiation, neonatal adaptation, and maternal clinical recovery.
  Interventions: Behavioral: ERAS Protocol
- Standard Perioperative Care (Active Comparator): Participants in this arm will receive standard perioperative care for cesarean delivery, which includes routine preoperative preparation, conventional intraoperative anesthesia and analgesia, standard postoperative monitoring, and usual mobilization and oral intake schedules. Skin-to-skin contact and breastfeeding initiation will be performed according to standard hospital practice, without additional ERAS-specific interventions. Outcomes include mother-infant and father-infant bonding, maternal postpartum depression, breastfeeding initiation, neonatal adaptation, and maternal clinical recovery.
  Interventions: Behavioral: Standard Perioperative Care

INTERVENTIONS:
Behavioral: ERAS Protocol — The Enhanced Recovery After Cesarean (ERAS) protocol includes shortened preoperative fasting, preoperative carbohydrate loading, multimodal opioid-sparing analgesia, early oral intake, early ambulation, and early removal of urinary catheter. The protocol also incorporates immediate or early skin-to-skin contact, early initiation of breastfeeding, and structured parental involvement. ERAS aims to optimize maternal postoperative recovery, reduce analgesic requirements, enhance mobility, improve patient satisfaction, and support early maternal-infant and paternal-infant bonding. No surgical technique is altered; only perioperative care differs from usual practice.
  Arms: ERAS Protocol
Behavioral: Standard Perioperative Care — Standard perioperative cesarean care includes routine preoperative fasting, no carbohydrate loading, conventional postoperative analgesia, delayed oral intake, delayed ambulation, and routine timing of urinary catheter removal. Immediate skin-to-skin contact and early breastfeeding are not systematically implemented. This arm reflects current institutional usual care and serves as the comparator to the ERAS protocol. No deviation from standard surgical or anesthetic techniques is introduced.
  Arms: Standard Perioperative Care

SUMMARY:
This is a multicenter, 1:1 parallel-group, randomized controlled trial designed to compare the effect of the Enhanced Recovery After Cesarean (ERAS) protocol versus standard perioperative care on mother-infant and father-infant bonding in women undergoing cesarean delivery. The study will initially be conducted as a single-center trial at Istanbul Okan University Hospital. Once adequate site preparation is completed, additional centers will be added to expand the study to a multicenter setting.

Primary Outcome:

The primary outcome is the total score on the Postpartum Bonding Questionnaire (PBQ) assessed on postpartum day 7, reflecting mother-infant bonding.

Secondary Outcomes:

Secondary outcomes include:

Maternal/Parental Postnatal Attachment Scale (MIBS) score at 2 hours postpartum (mother)

PBQ score at 24 hours postpartum (mother)

PBQ score at day 4 postpartum (mother)

PBQ score at day 7 postpartum (father-infant bonding)

Edinburgh Postnatal Depression Scale (EPDS) scores for mothers at 2 hours and 7 days postpartum

Time to initiation of breastfeeding

Requirement for neonatal intensive care unit (NICU) admission

Sample Size:

The total multicenter target sample size is n=300, with 150 participants in the ERAS group and 150 in the standard care group. The initial single-center phase at Okan University Hospital will enroll a target of n=100 participants (50 per group).

Randomization:

Participants will be randomized using a block and stratified randomization approach based on parity (primiparous vs multiparous) and planned type of anesthesia.

Blinding (Masking):

Due to the nature of the intervention, care providers cannot be blinded to group assignment. However, outcome assessors and data analysts will remain blinded to treatment allocation to minimize bias.

Study Timeline and Visits:

Participants will be evaluated at multiple time points following cesarean delivery: 2 hours postpartum, 24 hours postpartum, day 4 postpartum, and day 7 postpartum. All primary and secondary outcomes will be collected at the specified time points.

Significance and Rationale:

The ERAS protocol for cesarean delivery is designed to optimize perioperative care, enhance recovery, and potentially improve early parent-infant bonding. While previous studies have focused on maternal recovery and clinical outcomes, evidence regarding the impact of ERAS on both mother-infant and father-infant bonding remains limited. This trial aims to provide high-quality evidence on whether ERAS implementation can improve early bonding experiences, maternal mental health, breastfeeding initiation, and neonatal outcomes compared with standard perioperative care. The findings may guide future clinical practice and contribute to optimizing family-centered care in cesarean deliveries.

Key Features:

Multicenter, randomized controlled design

Parallel 1:1 allocation

Stratified randomization by parity and anesthesia type

Blinded outcome assessment and data analysis

Multiple postpartum evaluation points

Focus on psychosocial and clinical outcomes

Expected Contributions:

This study will provide comprehensive data on the feasibility and effectiveness of ERAS protocols in cesarean deliveries and their potential benefits for both maternal and paternal bonding with the newborn. The inclusion of both mother-infant and father-infant outcomes, as well as maternal mental health and breastfeeding indicators, ensures a holistic assessment of early family-centered outcomes.

DETAILED DESCRIPTION:
RATIONALE AND OBJECTIVES Introduction and Study Rationale

Cesarean delivery rates are increasing worldwide and in Turkey, highlighting the importance of not only physical recovery but also psychological and emotional recovery after birth. The Enhanced Recovery After Surgery (ERAS) protocol, initially developed for colorectal surgery, has recently been adapted to obstetrics as "ERAS for Cesarean." ERAS protocols offer concrete clinical benefits in the perioperative period, including enhanced patient comfort, reduced opioid use, earlier mobilization, and shortened hospital stay .

However, evidence regarding the effects of ERAS protocols on mother-infant bonding, breastfeeding success, and postpartum mental health in cesarean deliveries remains limited. Early contact between mother and infant during the first postpartum days increases oxytocin release, supporting not only uterine involution but also emotional bonding. Early skin-to-skin contact and early breastfeeding initiation reduce the risk of postpartum depression, while excessive opioid use and prolonged postoperative immobilization may negatively impact this process.

Key components of ERAS-including preoperative patient education and anxiety reduction, intraoperative multimodal analgesia, early oral intake, early mobilization, and early removal of Foley catheters-not only accelerate maternal physical recovery but may also enhance psychosocial recovery and parent-infant bonding. Recent pilot studies have reported that ERAS improves maternal satisfaction with birth experience, perceived self-efficacy, and reduces depressive symptoms. However, most of these studies were single-center, small sample size, and assessed psychosocial outcomes as secondary endpoints.

In Turkey, no randomized controlled trial has evaluated the relationship between ERAS protocols and parent-infant bonding after cesarean delivery. Moreover, father-infant bonding is an understudied area in obstetric literature. Cesarean delivery may limit fathers' initial contact with the newborn, potentially delaying emotional bonding. The ERAS protocol, by facilitating early skin-to-skin contact and integrating fathers into postpartum care, may mitigate these limitations.

This study aims, for the first time in Turkey, to evaluate the effects of the ERAS protocol on mother-infant and father-infant bonding using a multicenter, randomized controlled design. Findings will contribute to the literature on psychosocial outcomes of obstetric ERAS protocols and promote a holistic approach to postpartum recovery.

Primary Objective

The primary objective of this study is to evaluate the effect of the ERAS protocol, compared with standard perioperative care, on mother-infant bonding in women undergoing cesarean delivery. The primary endpoint will be the total score on the Postpartum Bonding Questionnaire (PBQ) measured on postpartum day 7. This will determine whether ERAS improves not only physical recovery but also emotional recovery and parent-infant bonding.

Secondary Objectives

Secondary objectives include:

Assessing the effect of ERAS on father-infant bonding at postpartum day 7 using the PBQ.

Evaluating early postpartum mother-infant bonding scores (MIBS at 2 hours, PBQ at 24 hours, day 4, and day 7).

Assessing the impact of ERAS on maternal postpartum depression using the Edinburgh Postnatal Depression Scale (EPDS) at 2 hours and day 7.

Investigating the effects of ERAS on time to first breastfeeding, breastfeeding success, and duration of skin-to-skin contact.

Evaluating neonatal outcomes, including NICU requirement, Apgar scores, and postpartum stabilization time.

Assessing maternal clinical recovery outcomes, such as early mobilization, oral intake, analgesic requirements, and length of hospital stay.

Evaluating maternal satisfaction with birth experience and perceived self-efficacy following ERAS implementation.

3. HYPOTHESES

Mothers receiving the ERAS protocol will have significantly higher mother-infant bonding scores (PBQ total) on postpartum day 7 compared with those receiving standard care.

Fathers in the ERAS group will demonstrate higher father-infant PBQ scores on postpartum day 7 than fathers in the standard care group.

ERAS will increase early postpartum mother-infant bonding (MIBS score at 2 hours) and reduce postpartum depression scores (EPDS).

ERAS implementation will shorten time to first breastfeeding, extend duration of skin-to-skin contact, and improve breastfeeding success.

Neonatal outcomes, including Apgar scores, NICU admission rates, and postpartum adaptation, will be improved in the ERAS group compared with standard care.

Maternal clinical recovery indicators-including early mobilization, oral intake, analgesic requirement, and hospital stay-will be superior in the ERAS group.

ERAS will enhance maternal satisfaction with birth experience and perceived self-efficacy.

ELIGIBILITY:
IInclusion Criteria:

Pregnant women aged 18-60 years.

Singleton, live fetus, and ≥37 weeks of gestation.

Undergoing elective or medically indicated cesarean delivery.

Ability to read and understand Turkish (for questionnaire validity).

Mothers and fathers willing and able to complete postpartum follow-up assessments (2 hours, 24 hours, day 4, day 7).

Provision of written informed consent by mother and, if participating, by father/partner.

Maternal postpartum clinical stability (no condition precluding questionnaire completion).

❌ Exclusion Criteria (Dışlanma Kriterleri)

Exclusion Criteria:

Preterm birth (<37 weeks) or multiple gestation (twins, triplets).

Stillbirth, early neonatal death, or major congenital anomaly.

Newborn requiring prolonged NICU stay preventing bonding assessments.

Maternal severe obstetric complications:

Massive postpartum hemorrhage

Hysterectomy

Severe preeclampsia or eclampsia

Severe postpartum infection

Maternal active psychiatric disorder or use of psychotropic medication.

Maternal need for high-dose opioid analgesia or sedation interfering with bonding assessments.

Inability to read/understand Turkish or cognitive impairment preventing questionnaire completion.

Failure to complete follow-up visits (2 hours, 24 hours, day 4, day 7).

Withdrawal of consent at any time.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Estimated)
Dates: Start 2025-12-13 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Mother-Infant Bonding Score at Postpartum Day 7 (PBQ Total Score) | Postpartum Day 7
  The primary outcome is the maternal bonding score assessed on postpartum day 7 using the validated Postpartum Bonding Questionnaire (PBQ). The PBQ total score evaluates the quality of early emotional bonding between mother and infant across domains including affection, rejection, and anxiety. Higher scores indicate better bonding. The ERAS protocol is hypothesized to improve bonding through enhanced maternal recovery, reduced postoperative discomfort, earlier mobilization, improved emotional well-being, and structured support for early skin-to-skin contact and breastfeeding. PBQ is administered by trained staff blinded to group allocation.

SECONDARY OUTCOMES:
Mother-Infant Bonding Score at 2 Hours Postpartum (MIBS Score) | 2 hours postpartum
  Early maternal bonding is assessed using the validated Mother-to-Infant Bonding Scale (MIBS) at 2 hours postpartum. The scale evaluates emotional response, closeness, and early attachment behaviors. Higher scores indicate better bonding. Trained assessors blinded to group allocation administer the scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Okan University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ituk U, Habib AS. Enhanced recovery after cesarean delivery. F1000Res. 2018 Apr 27;7:F1000 Faculty Rev-513. doi: 10.12688/f1000research.13895.1. eCollection 2018. PMID 29770203
- [Result] Ozdemir MG, Gunaydin B, Bayram M, Hirfanoglu IM. Effect of enhanced recovery after surgery (ERAS) protocol on maternal and fetal outcomes following elective cesarean section: an observational trial. BMC Pregnancy Childbirth. 2025 Apr 29;25(1):517. doi: 10.1186/s12884-025-07583-3. PMID 40301800
- [Result] Widstrom AM, Brimdyr K, Svensson K, Cadwell K, Nissen E. Skin-to-skin contact the first hour after birth, underlying implications and clinical practice. Acta Paediatr. 2019 Jul;108(7):1192-1204. doi: 10.1111/apa.14754. Epub 2019 Mar 13. PMID 30762247
- [Result] Bigelow A, Power M, MacLellan-Peters J, Alex M, McDonald C. Effect of mother/infant skin-to-skin contact on postpartum depressive symptoms and maternal physiological stress. J Obstet Gynecol Neonatal Nurs. 2012 May-Jun;41(3):369-82. doi: 10.1111/j.1552-6909.2012.01350.x. Epub 2012 Apr 26. PMID 22537390
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/29770203/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40301800/

DOCUMENTS (4):
  • Study Protocol (2025-11-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT07276126/Prot_000.pdf
  • Statistical Analysis Plan (2025-11-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT07276126/SAP_001.pdf
  • Informed Consent Form: INFORMED CONSENT FORM - MOTHER (2025-11-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT07276126/ICF_002.pdf
  • Informed Consent Form: INFORMED CONSENT FORM - FATHER (2025-11-04): https://cdn.clinicaltrials.gov/large-docs/26/NCT07276126/ICF_003.pdf